CLINICAL TRIAL: NCT03327129
Title: Identifying the Neural Basis of Capability for Suicide
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: SRO-01
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Suicide; Suicidal Ideation; Psychiatric Illness
MeSH Terms: conditions — Depressive Disorder, Major; Suicide; Suicidal Ideation; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — A urine sample to test for toxicology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Subjects will have no personal or family psychiatric history and no suicide attempts.
  Interventions: Procedure: fMRI
- Patients with SI: Subjects will have suicidal ideation (Hamilton Depression Rating Scale suicide item >=2).
  Interventions: Procedure: fMRI

INTERVENTIONS:
Procedure: fMRI — An fMRI scan will be conducted to collect neuroimaging data. The scanning session will consist of a structural MRI, followed by resting state and task-based functional MRI protocol.

SUMMARY:
Since capability for suicide involves overriding potential pain, and the opioid system plays a strong role in controlling pain perception, it follows that capability for suicide may be impacted by the opioid system. The goal of the proposed research is to identify the neural network underlying capability for suicide in order to determine if it can be a target for identifying high-risk individuals and for intervention.

DETAILED DESCRIPTION:
Little evidence exists distinguishing individuals with suicidal ideation (SI) from those at risk for suicidal behaviour, illustrating the need for more comprehensive biomarkers for clinicians to guide their treatment approach and for new treatment avenues. Current theories of suicide have suggested the importance of an individual's capability for suicide in predicting suicide attempt or death. Building on this, Yovell and colleagues (2016) provided important preliminary data that the opioid system affects suicide risk, but the neural mechanisms and their relationship to capability for suicide are unclear. The goal of the proposed research is to identify the neural network underlying capability for suicide using functional magnetic resonance imaging (fMRI) in order to determine if it can be a target for identifying high-risk individuals and for intervention.

ELIGIBILITY:
Inclusion criteria for patients:

* Age between 18-70
* Capability of giving informed consent
* Not currently pregnant or lactating (due to potential confounding of brain activity as a result of differing hormone levels)

Exclusion criteria for patients:

* Lifetime history of any substance abuse, psychosis
* Current use of any opioid acting drugs
* Current use of any prescription pain medication
* Use of over the counter pain medications within 15 hours of brain scan
* For daily users of a benzodiazepine, stimulant or atypical antipsychotic, dose within 12 hours of brain scan
* For as needed users of a benzodiazepine, stimulant or atypical antipsychotic, dose within 2 weeks of brain scan. This is because non-daily use will have more unpredictable effects on brain imaging results than those who are using these medications on a regular basis. The 2 weeks will ensure the drug is not in the system.
* Medical condition requiring immediate investigation or treatment
* Participation in experimental treatment trials for the study duration.

Healthy control inclusion criteria: Ages between 18 and 70 years, capable of giving informed consent, not pregnant or lactating, no lifetime history of Axis I/II disorders, no history of antidepressant or mood stabilizer use, no treatment for acute or ongoing medical condition, no use of any over the counter pain medication for at least 15 hours prior to the brain scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will recruited from Mental Health Clinics at St. Michael's Hospital from Mood Disorders Clinics and self-referrals from advertisements in Mental Health Department.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Neural network underlying acquired capability for suicide | 2 weeks
  Measure the correlation between acquired capability for suicide and brain activity during a pressure pain task using fMRI in patients

SECONDARY OUTCOMES:
Correlation between pain task performance and acquired capability for suicide | 2 weeks
  Assess the association between pain task ratings and acquired capability for suicide in patients

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada